CLINICAL TRIAL: NCT01232634
Title: External Validation of Ultrasound as a Diagnostic Tool for Assessment of Hemophilic Arthropathy of Knees and Ankles. MRI Correlation.
Brief Title: Validation of Ultrasound as a Diagnostic Tool for Assessment of Hemophilic Arthropathy of Knees and Ankles
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University of Sao Paulo (Other); Federal University of São Paulo (Other); University of Campinas, Brazil (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Andrea Doria, Clinician Scientist, The Hospital for Sick Children
Other Study IDs: 1000010841
Record Dates: First submitted 2010-10-29; First posted 2010-11-02 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Hemophilia; Hemophilic Arthropathy
Keywords: pediatrics; haemophilia; ultrasound; MRI; arthropathy
MeSH Terms: conditions — Hemophilia A; Joint Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Subjects

SUMMARY:
The purpose of this study is to test the external validity of the systemic ultrasound protocol for data acquisition and interpretation, in order to diagnose soft tissue and osteochondral abnormalities in hemophilic children.

DETAILED DESCRIPTION:
Ultrasound has advantages over MRI as it is less expensive, does not require sedation and is more readily available in centres around the world. Given these characteristics of ultrasound it is an ideal imaging tool for early assessment of hemophilic joints in countries whose access to MRI is limited. Early evaluation of soft tissue changes in young hemophilic patients may lead to earlier interventions and better mid-term and long-term clinical outcomes. By this way the joint function of hemophilic patients can be preserved, saving their joints from severe arthropathy and offering them the possibility of a normal professional life in the society.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A (factor VIII deficiency ≤1%) or B (factor IX deficiency ≤1.0%)
* Cooperative patients (age of 7 to 18 years old)
* Patients under 7 years old who have clinical evidence of arthropathy and imaging studies are required for clinical reasons. In these cases, the procedures may be done under sedation.
* Male sex (higher prevalence in males)
* History of previous ankle or knee bleed

Exclusion Criteria:

* Co-morbid illness such as juvenile idiopathic arthritis, muscular dystrophy, neuropathic arthropathy that cause osteoarticular findings that may obscure or confound the hemophilia-based joint findings
* Non-cooperative patients
* Active bleed (defined as evidence of a recent bleed with one week of the proposing imaging studies and/or musculoskeletal changes on physical examination suggestive of a bleed within one week of the proposed imaging studies).
* Prior synovectomy

Ages: 7 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children attending the Hemophilia clinics at the participating institutions (Universidade de São Paulo, Universidade Federal de São Paulo and Universidade Estadual de Campinas), who have a history of ankle or knee bleed(s), will be recruited to take part in this study.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Ultrasound findings according to the International Prophylaxis Study Group (IPSG) scale | Day 1
  The readers will mark all the positive findings on a standardized spreadsheet and providing a final score for each component of the scale. Color Doppler findings will be rated as normal (grade 0), mild/moderate (grade 1) or severe (grade 2) synovial hyperemia according to an atlas that shows the intensity of hyperemia, which has been prepared by our group.

SECONDARY OUTCOMES:
MRI findings according to the International Prophylaxis Study Group (IPSG) scale | Day 1
  The readers will interpret the MRI findings in an additive way, i.e., marking all positive findings on a standardized spreadsheet and providing a final score for the soft tissue and osteochondral components of the MRI scale.
X-ray findings according to the Pettersson radiographic system | Day 1
  Each joint will be rated on a 13-point score after the Pettersson system.
Physical Assessment according to the HJHS and FISH scores | Day 1
  Each knee, elbow and ankle joint receives a numeric score, which can be compared to itself over time to determine whether it is showing degeneration due to bleeding. FISH score is a seven item measure of disability used to evaluate change in functional independence over time.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Doria, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (4):
- Brazil (3):
  - Universidade de Sao Paulo, São Paulo
  - Universidade Estaduale de Campinas, São Paulo
  - Universidade Federal de Sao Paulo, São Paulo
- The Hospital for Sick Children, Toronto, Ontario, Canada